CLINICAL TRIAL: NCT03149718
Title: Prescription Opioid Misuse: Pharmacist-Delivered Intervention at Point of Service
Brief Title: Community Pharmacists and Opioid Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jerry Cochran, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17010410; R21DA043735 (NIH)
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Opioid Misuse
Keywords: Pharmacy; Intervention; Medication Adherence
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMC (n=23) (Active Comparator): Standard Medication Counseling.
  Interventions: Behavioral: Standard Medication Counseling (SMC)
- BI-MTM (n=23) (Experimental): Brief Intervention Medication Therapy Management.
  Interventions: Behavioral: Brief Intervention Medication Therapy Management

INTERVENTIONS:
Behavioral: Brief Intervention Medication Therapy Management — BI-MTM is designed to: (1) eliminate opioid medication misuse, (2) promote opioid regimen adherence, (3) connect participants with Patient Navigation to increase patient self-management activation for health conditions that increase risk for misuse (Patient Navigation is an evidence-based chronic care intervention), and (4) provide naloxone rescue training referrals.
  Arms: BI-MTM (n=23)
Behavioral: Standard Medication Counseling (SMC) — Standard Medication Counseling (SMC; n=23; i.e., treatment-as-usual condition). Standard Medication Counseling is the Centers for Medicaid and Medicare Services requirement for pharmacists in the US wherein pharmacy patients filling prescriptions receive information and opt-in counseling.
  Arms: SMC (n=23)

SUMMARY:
Opioid medication misuse and overdose have reached epidemic proportions in the US. Community pharmacy is a potentially valuable resource for addressing opioid medication misuse. This study will manualize and establish the feasibility, acceptability, and clinical effect of a community pharmacist-led intervention aimed at: improving opioid mediation regimen adherence, eliminating misuse, connecting patients to additional care, and safeguarding against overdose.

DETAILED DESCRIPTION:
The current small scale single-blinded randomized controlled study will build on our preliminary studies by manualizing and examining the feasibility, acceptability, and clinical effect for the Brief Intervention Medication Therapy Management (BI-MTM) model. BI-MTM is a multicomponent community pharmacy-based intervention. BI-MTM is designed to: (1) promote opioid medication regimen adherence, (2) reduce opioid medication misuse, (3) connect participants with patient navigation (a chronic condition care model) to increase self-management of health conditions that increase risk for misuse, and (4) provide naloxone rescue training referrals. Patients will be screened across 14 months for opioid medication misuse in an urban community pharmacy affiliated with a major medical system. Patients positive for misuse will be randomly assigned to BI-MTM (n=23) or Standard Medication Counseling (n=23). Standard Medication Counseling is the Centers for Medicaid and Medicare Services requirement for pharmacists in the US wherein pharmacy patients filling prescriptions receive information and opt-in counseling. This study will demonstrate feasibility and acceptability of BI-MTM for community pharmacy patients who misuse their opioid medications for future intervention implementation in a fully powered randomized trial. This study will also generate preliminary data regarding opioid medication misuse elimination and increases in participant self-management activation for comorbid health conditions that increase risk for misuse.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Misuse

  -≥18 years
* English speaking

Exclusion Criteria:

* Are pregnant (given potential pre/post-natal opioid use complications among pregnant women/offspring)
* Cannot provide collateral contact information for ≥2 contact persons (to ensure consistent contact/follow up)
* Do not have a reliable landline or mobile phone to be contacted by study staff
* Are only filling buprenorphine (given some formulations are not indicated for pain)
* Plan to leave the area for an extended period of time in the next 3 months
* Have had a psychotic and/or manic episode in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | Month 21 of Study
  Intervention feasibility will be established through delivery of all BI-MTM components to 85% of BI-MTM recipients.
Intervention acceptability | Month 21 of Study
  Intervention acceptability will be demonstrated though qualitative interviews.

SECONDARY OUTCOMES:
Opioid Misuse | Month 21 of Study
  Opioid misuse will be demonstrated by the Prescription Opioid Misuse Index (POMI).
Patient Self-Management | Month 21 of Study
  Patient self-management activation misuse than will be captured by the Patient Activation Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Cochran, Ph.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Falk Pharmacy, Pittsburgh, Pennsylvania
  - Medicine Shoppe, Somerset, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided